CLINICAL TRIAL: NCT06481254
Title: Effect of Hawthorn Vinegar, Black Mulberry Syrup and Green Tea on Quality of Life Related to Oral Mucositis and Oral Health in Individuals With Diabetes: Single Blind Randomized Controlled Study
Brief Title: Effect of Hawthorn Vinegar, Black Mulberry Syrup and Green Tea on Oral Mucositis
Acronym: Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Bayburt University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Assistant professor, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS06022024
Record Dates: First submitted 2024-06-23; First posted 2024-07-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Mucositis; Quality of Life
Keywords: Hawthorn vinegar; Black mulberry syrup; Mucositis; Green tea; Quality of life.
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Intervention Model Description: The sample size of the study was calculated as 128 individuals in total (32 for each group) for 4 groups (hawthorn vinegar, black mulberry syrup, green tea, control group) with an effect size of 0.25 with α=0.05 and the power of the targeted test was 0.80 (80%) in the G*Power 3.1.9.7 program, which could not be used as a reference since there was no previous four-group study on the subject. Each group was increased to account for drop-outs and deaths and a total of 140 individuals, 35 for each group, were included in the study
Who Masked: Investigator
Masking Description: The principal investigator completed the consent and assent forms after explaining the purpose of the study to all participants. In the research planned as a single-blind randomized controlled clinical study, the other researcher who applied the data collection tools to reduce bias was not told who the experimental groups (hawthorn vinegar group, black mulberry syrup group, green tea group) and the patients with DM in the control group were.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hawthorn Vinegar Group (Experimental): Before starting the study (pre-test/0. week), "Patient Information Form", "OAG" and "OHQoL-UK" were administered to all group participants to evaluate the level of oral mucositis in patients. In addition to routine oral mucositis treatment, patients with DM in the hawthorn vinegar group gargled with 1 tablespoon (10 cc) of diluted hawthorn vinegar (mixed with 40 cc water) for 1 minute 15-20 minutes before meals 3 times a day for 14 days. "OAG" and "OHQoL-UK" were administered again on the 7th day (interim-measurement) and 14th day/end of the study (post-test).
  Interventions: Other: Hawthorn Vinegar Group
- Black Mulberry Syrup Group (Experimental): Before starting the study (pre-test/0. week), "Patient Information Form", "OAG" and "OHQoL-UK" were administered to all group participants to evaluate the level of oral mucositis in patients. In addition to routine oral mucositis treatment, patients with DM in the black mulberry syrup group gargled with 1 tablespoon (10 cc) of pure black mulberry syrup for 1 minute 15-20 minutes before meals 3 times a day for 14 days. "OAG" and "OHQoL-UK" were administered again on the 7th day (interim-measurement) and 14th day/end of the study (post-test).
  Interventions: Other: Black Mulberry Syrup Group
- Green Tea Group (Experimental): Before starting the study (pre-test/0. week), "Patient Information Form", "OAG" and "OHQoL-UK" were administered to all group participants to evaluate the level of oral mucositis in patients. In addition to routine oral mucositis treatment, patients with DM in the green tea group gargled with 50 cc green tea for 1 minute 15-20 minutes before meals 3 times a day for 14 days. "OAG" and "OHQoL-UK" were administered again on the 7th day (interim-measurement) and 14th day/end of the study (post-test).
  Interventions: Other: Green Tea Group
- Control Group (No Intervention): Patients in the control group received no any treatment other than routine oral mucositis treatment and data collection tools. "Patient Information Form", "OAG" and "OHQoL-UK" were administered to the patients before the study (pre-test/0th week) and "OAG" and "OHQoL-UK" were administered again on the 7th day (mid-measurement) and 14th day/end of the study (post-test).

INTERVENTIONS:
Other: Hawthorn Vinegar Group — To routine oral mucositis treatment, patients with DM in the hawthorn vinegar group gargled with 1 tablespoon (10 cc) of diluted hawthorn vinegar (mixed with 40 cc water) for 1 minute 15-20 minutes before meals 3 times a day for 14 days.
  Arms: Hawthorn Vinegar Group
Other: Black Mulberry Syrup Group — To routine oral mucositis treatment, patients with DM in the black mulberry syrup group pure black mulberry syrup for 1 minute 15-20 minutes before meals 3 times a day for 14 days.
  Arms: Black Mulberry Syrup Group
Other: Green Tea Group — To routine oral mucositis treatment, patients with DM in the green tea group gargled with 50 cc green tea for 1 minute 15-20 minutes before meals 3 times a day for 14 days.
  Arms: Green Tea Group

SUMMARY:
In this context, this study investigated the quality of life related to oral mucositis and oral health in patients with DM using hawthorn vinegar, black mulberry syrup and green tea.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic metabolic disease that causes serious damage to the heart, blood vessels, eyes, kidneys and nerves. Both the number of cases and the prevalence of diabetes have been increased rapidly over the past 30 years. According to the report of the International Diabetes Federation (IDF) Report, approximately 537 million people worldwide (700 million in 4045) have diabetes and 6.5 million people were reported to have died due to diabetes in 2021. In Turkey, it is estimated that approximately 9 million people (about 13.5 million in 2045) are diagnosed with diabetes and approximately 80 thousand people will die from diabetes.

Prolonged hyperglycemia in DM can lead to microvascular (nephropathy, retinopathy and neuropathy) and macrovascular (peripheral vascular disease, hypertension, cerebrovascular disease, ischaemic heart disease) complications. However, due to poorly controlled DM, complications can be seen in the oral mucosa of patients with many immunological and metabolic changes. Oral complications seen in patients with DM include hyposalivation, xerostomia, bacterial, viral and fungal infections, poor wound healing, increased severity and incidence of caries, gingivitis and periodontal disease, periapical abscess, and burning mouth syndrome (BMS). These complications can lead to the development of oral mucositis in patients.

Many pharmacological and non-pharmacological agents are used in the prevention/treatment of oral mucositis. According to the classification of the National Center for Complementary and Integrative Health (NCCAM), complementary therapies methods are divided into three groups as nutritional, psychological and physiological and other complementary approaches. However, it is reported in the literature that complementary therapies such as cryotherapy (oral cooling), honey, propolis, vitamin E, selenium, aloe vera, black mulberry, apple cider vinegar, rose water and green tea are effective in the treatment of oral mucositis. Again in the literature, there are studies in which the effect of black mulberry syrup in patients with Chronic Obstructive Pulmonary Disease (COPD), apple cider vinegar and rose water mixture in cancer patients and green tea in the treatment of oral mucositis has been proven.

Oral mucositis is one of the oral diseases that can cause oral dysfunction, dysphagia and reduced oral health-related quality of life in patients. Oral and dental health affects a person's quality of life by affecting their physiological, psychological and social functioning. However, improving oral health is part of nursing care. In order to maintain a good quality of life, it is necessary to improve awareness of oral complications that occur in patients with DM. In the literature reviewed, only one experimental study was found in cancer patients in which oral mucositis-related quality of life was evaluated. There is no international or Turkish study on the treatment of oral mucositis in patients with DM. There are also no studies comparing hawthorn vinegar, black mulberry syrup and green tea in different sample groups. In this context, this study investigated the quality of life related to oral mucositis and oral health in patients with DM using hawthorn vinegar, black mulberry syrup and green tea.

ELIGIBILITY:
Inclusion Criteria:

* Overs 18 years of age,
* Voluntary participation in the study,
* Be lucid and able to communicate,
* Be diagnosed with DM for at least 3 months ago,
* Willing to use either hawthorn vinegar, black mulberry syrup or green tea as a complementary treatment for oral mucositis,
* HbA1c ≥ 7% (Wang and Hng, 2021),
* Oral mucositis score of 14< in oral assessment.

Exclusion Criteria:

* Having a known psychological disorder,
* Having HbA1c <7%,
* Not having oral mucositis,
* Having hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Oral Assessment Guide (OAG) | 14 Days
  The "OAG" is useful for assessing and recording the individual's daily oral condition, as well as detecting the presence of mucositis and evaluating the effectiveness of treatment. The "OAG" consists of 8 categories including voice, dysphagia, lips, tongue, saliva, mucous membranes, gums and teeth/prostheses.
  "OAG" was administered again on the 7th day (interim-measurement) and 14th day/end of the study (post-test).
Oral Health Related Quality of Life Scale (OHQoL-UK) | 14 Days
  The 5-point Likert-type scale, which consists of a total of 16 items to determine the degree of impact of teeth, gums, mouth or prosthesis, consists of 4 dimensions: "symptom" (items 1-2), "physical condition" (items 3-7), "psychological condition" (items 8-12) and "social condition" (items 13-16). Each item in the scale is scored as "Very bad effect-1, bad effect-2, no effect-3, good effect-4, very good effect-5". The total score of the scale varies between 16-80, and a high score indicates a high level of oral and dental health-related quality of life. The Cronbach alpha value of the scale was reported as 0.94.
  "OHQoL-UK" was administered again on the 7th day (interim-measurement) and 14th day/end of the study (post-test).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Demirağ, Dr.Öğr.Üyesi, Principal Investigator — Study Principal Investigator Gümüşhane Universıty
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No